CLINICAL TRIAL: NCT01218282
Title: Different Methods of Home Exercise Training in COPD Patients
Brief Title: Exercise Training in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Annalisa Cogo, University of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ExTCOPD01
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: COPD
Keywords: COPD; home exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Home Exercise Training Group A1 (Experimental): Patients assigned to this arm maintain the prescribed walking speed during the training with a metronome
  Interventions: Behavioral: Home exercise training
- Home Exercise Training Group A2 (Experimental): Patients assigned to this arm cover a fixed distance in a given period of time.
  Interventions: Behavioral: Home exercise training
- Control (No Intervention)
  Interventions: Behavioral: NO Exercise Training

INTERVENTIONS:
Behavioral: Home exercise training — 20-30 min/day for at least 4 days/week
  Other Names: Pulmonary Rehabilitation
  Arms: Home Exercise Training Group A1; Home Exercise Training Group A2
Behavioral: NO Exercise Training — No intervention
  Other Names: No intervention
  Arms: Control

SUMMARY:
Exercise training is the key component of respiratory rehabilitation.The success of long-term program resides in the integration between exercise prescription and patients'compliance with home training. This can be difficult for patients, especially in terms of understanding the exercise intensity.

This study is designed to evaluate different methods of exercise training at home, to help understanding and maintaining the walking intensity in COPD patients. Outcome: exercise performance, daily physical activity and respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients. All patients are at stable state, free from an exacerbation from at least 3 months.

Exclusion Criteria:

* COPD patients with a recent history of cardiovascular disease and other diseases that would interfere with exercise performance.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Cogo, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Pulmonary respiratory unit- University Hospital, Ferrara, Ferrara, Italy